CLINICAL TRIAL: NCT03657823
Title: Fetal Growth and Pregnancy Complications Among Women With Heart Disease in Norway: a Cohort Study
Brief Title: Fetal Growth and Pregnancy Complications Among Women With Heart Disease
Acronym: PreCor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ingvil Krarup Sørbye, Consultant OBGYN, MD PhD, Oslo University Hospital
Other Study IDs: 2018/414
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Congenital Heart Disease; Pregnancy Complications; Arrhythmias, Cardiac; Hypertension in Pregnancy
MeSH Terms: conditions — Heart Defects, Congenital; Pregnancy Complications; Arrhythmias, Cardiac; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples Without DNA — Biomarkers in maternal serum iin subgroups

GROUPS / COHORTS (2):
- Fetal growth cohort: Longitudinal measurements of fetal growth, fetal circulation and maternal circulation
- Hypertensive cohort: Retrospective cohort of women with heart disease that underwent oregnancy and childbirth

SUMMARY:
An increasing proportion of women with heart disease now go through pregnancy and childbirth. More knowledge about the risk of complications and adverse outcomes for the mother and the baby is needed to guide clinical care in this diverse patient group.

The purpose of this study is to, in a cohort of pregnant women with heart disease;

* determine fetal growth, and risk of fetal growth restriction and preterm birth
* determine whether maternal blood biomarkers are associated with development of preeclampsia, the time of delivery and maternal and perinatal adverse outcomes
* determine the risk of hypertensive pregnancy complications

The expected outcome of the project is to increase the knowledge of optimal diagnosis and treatment of women with heart disease that go through pregnancy to be able to improve clinical care and the outcomes for mother and baby.

DETAILED DESCRIPTION:
Heart disease is about to become the most important cause of maternal deaths in industrialized countries. In addition, heart disease in pregnancy is associated to an increased rate of fetal growth restriction, premature birth, preeclampsia and other pregnancy complications for the mother and the baby. As many women with congenital or acquired heart disease now go through pregnancy and childbirth, more knowledge about the risk of complications and adverse outcomes for the mother and the baby is needed to guide clinical care in this diverse patient group.

The National Unit for Pregnancy and Heart Disease is located at Oslo University Hospital, Rikshospitalet, and receive moderate and high risk pregnant women as referrals from hospitals nationwide for follow-up and treatment. The unit has established Oslo University Hospital Register for Pregnancy and Heart disease; a quality register for maternal and fetal outcome in women with heart disease.

The purpose of this study was therefore to, in a cohort of pregnant women with heart disease;

* determine fetal growth, and risk of fetal growth restriction and preterm birth
* determine whether maternal blood biomarkers are associated with development of preeclampsia, the time of delivery and maternal and perinatal adverse outcomes
* determine the risk of hypertensive pregnancy complications

By the next two years, 150 patients will be included in two prospective longitudinal studies. In the first study fetal growth and utero-placental-fetal blood flow will be assessed by serial measurements at specific gestational ages. The mother's cardiac function will also be measured. Primary outcome is fetal growth curve and wellbeing at birth.

In the second study, biomarkers in maternal serum will be measured during the last half of pregnancy to assess if angiogenetic factors are prognostic for the risk of hypertensive complications.

In the last study the researchers will use retrospective data from the Oslo University Hospital Register for Pregnancy and Heart disease to determine the association between heart disease and hypertensive complications in a retrospective cohort of approximately 800 patients.

The expected outcome of the project is to increase the knowledge of optimal diagnosis and treatment of women with heart disease that go through pregnancy to be able to improve clinical care and the outcomes for mother and baby.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with heart disease before or during pregnancy classified as maternal WHO risk class 2-4

Exclusion Criteria:

* Non-consent

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with congenital or aquired heart disease that are enrolled or referred to Oslo University Hospital for follow-up in pregnancy and childbirth according to criteria set by the Norwegian National Treatment Unit for Heart Disease and Pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Fetal growth | From gestational week 12 until time of birth of baby
  Serial measurements of fetal biometry
Occurrence of hypertension/preeclampsia in pregnancy or postpartum | From time of study inclusion until time of discharge from maternity unit after birth of baby
  Diagnosis in index pregnancy or postpartum until discharge from maternity unit
Fetoplacental circulation | From gestational week 12 until time of birth of baby
  Serial measurements of fetoplacental circulation

CONTACTS AND LOCATIONS:
Overall Officials: Mette E Estensen, PhD, MD, Study Director — Oslo University Hospital, Dep. of Cardiology
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Upon individual application
Supporting Information: Study Protocol, SAP
Time Frame: After June 2021
Access Criteria: Upon individual application